CLINICAL TRIAL: NCT06189937
Title: Culturally Adapted Cognitive Behavioral Therapy to Reduce Psychological Distress of Individuals Affected by the Earthquake: A Pilot Randomized Controlled Trial
Brief Title: Group CA-CBT Intervention to Reduce Psychological Distress of Earthquake Survivors
Acronym: CARED-ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.060.IRB3.027
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-01

CONDITIONS: Psychological Distress; Depressive Symptoms; Well-Being, Psychological
Keywords: earthquake survivor; culturally adapted treatment; mental health; cognitive behavioral therapy
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A pilot randomized control trial involving 60 participants will be conducted. 30 randomly allocated participants will receive CA-CBT and 30 randomly allocated participants will receive Enhanced Care as Usual (E-CAU) as the control group. One week after the completion of the sessions, all participants including control group participants will have post-assessments consisting of the same questionnaires as baseline assessment with assessors. One month after the post-assessment, with the assessors, all participants including control group participants will have follow-up assessments consisting of the same questionnaires as baseline and post-assessments. After completing all assessments, CA-CBT will be offered to control group participants.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded to their study arm due to the nature of the intervention, but outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Culturally Adapted Cognitive Behavioral Therapy (CA-CBT) (Experimental): Participants in the experimental group will receive an 8-session group CA-CBT.
  Interventions: Behavioral: Culturally Adapted Cognitive Behavioral Therapy (CA-CBT)
- Enhanced Care as Usual (E-CAU) (No Intervention): Participants in the control group will receive pamphlets containing information on mental health issues following earthquakes, coping strategies, and free psychological support centers. After completing all assessments, CA-CBT will be offered to these participants.

INTERVENTIONS:
Behavioral: Culturally Adapted Cognitive Behavioral Therapy (CA-CBT) — In this study, an 8- session (90 to 120 minutes) group version of the transdiagnostic intervention CA-CBT tailored for earthquake survivors will be applied.
  Contents of the sessions are:
  1. Education on psychological trauma and its treatment, and basics of emotion regulation techniques
  2. Education on anxiety and depressive disorders and their treatment
  3. Muscle relaxation and stretching exercises
  4. Education about depressive and grief-related disorders and disturbing memories protocol
  5. Interoceptive exposure: head rotation and hyperventilation
  6. Anxiety, worry, and stress
  7. Anger and anger protocol; breathing exercises
  8. Somatic complaints, sleep disturbance, and closing
  There will be one facilitator and one co-facilitator. Groups will consist of 12-13 participants.
  Arms: Culturally Adapted Cognitive Behavioral Therapy (CA-CBT)

SUMMARY:
Earthquakes in Türkiye cause survivors to develop serious and prolonged mental health issues and adapted versions of cognitive behavioral therapy has proven to be successful in addressing these concerns.The main goal of this pilot randomized control trial (RCT) is to test potential effectiveness of Culturally Adapted Cognitive Behavioral Therapy (CA-CBT) in reducing psychological distress and depressive symptoms and increasing well-being of earthquake survivors.

DETAILED DESCRIPTION:
Türkiye was struck by two large earthquakes with moment magnitudes 7.7. and 7.6, on the 6th of February 2023. The disaster resulted in more than 50 thousand people losing their lives, more than 107 thousand people getting injured and more than 84 thousand buildings being demolished, severely damaged or slated for demolition. After the earthquakes, various mental health issues can emerge among the survivors such as depression, anxiety disorders, posttraumatic stress disorder, sleep problems, prolonged grief disorder, decrease in quality of life, increase in suicidality and substance use, and their effects can be prolonged if not treated.

An effective treatment method for the mental health issues that the earthquake survivors may experience is cognitive behavioral therapy (CBT) which is effective both in individual and group formats. Moreover, culturally adapted versions of CBT demonstrated higher effectiveness. One such adaptation, developed as a transdiagnostic intervention by Devon Hinton, is known as Culturally Adapted CBT (CA-CBT), which has shown effectiveness across various cultures and countries. It has been successfully applied to depressed and traumatized women in Türkiye, reducing depressive symptoms and PTSD. CA-CBT incorporates emotion regulation techniques, mindfulness and stretching exercises as well as cognitive-behavioral approach principles. Some advantages of the CA-CBT are: (1) as a transdiagnostic intervention, it can be applied to treat various psychopathologies (2) as a group intervention, it can be applied to multiple individuals simultaneously, (3) as an 8-session intervention, it can improve mental health in the short term.

CA-CBT has not been tested with a population specifically consisting of individuals affected by earthquakes before. This pilot randomized control trial (RCT) aims to assess the potential effectiveness and feasibility of CA-CBT, specifically tailored for the earthquake survivors, and their mental health issues following the disaster. The main research questions of the study are whether the group CA-CBT is effective in decreasing psychological distress and depressive symptoms and increasing well-being among earthquake survivors one month after post-assessment.

The study is planned to be conducted with the collaboration with non-governmental organizations giving services to earthquake survivors. After the baseline assessment, eligible 60 participants will be randomized to two arms according to the 1:1 principle with automatized randomization software. 30 randomly allocated participants will receive CA-CBT and 30 randomly allocated participants will receive Enhanced Care as Usual (E-CAU) as the control group. One week after the completion of the sessions, all participants including control group participants will have post-assessments consisting of the same questionnaires as baseline assessment. One month after the post-assessment, all participants including control group participants will have follow-up assessments consisting of the same questionnaires as baseline and post-assessments.

If CA-CBT proves effective for individuals affected by earthquakes, it can be disseminated among mental health care professionals. Consequently, more earthquake survivors can access this high-quality evidence-based intervention adapted to their culture.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older.
* Having experienced the earthquake.
* Having a considerable amount of psychological distress: scoring 16 or higher on the Kessler Psychological Distress Scale (K10).

Exclusion Criteria:

* Having a severe mental disorder (conducted by a trained assessor).
* Presenting suicidality (assessed by the Problem Management Plus Suicidality Tool).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Kessler Psychological Distress Scale (K-10) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  K-10 is a 10-item scale that measures psychological distress. Each item is scored from 1 (none of the time) to 5 (all of the time) and ranges between 10 and 50. Higher scores indicate higher levels of psychological distress.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  PHQ-9 is a 9-item questionnaire that measures depressive symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 27. Higher scores indicate higher depressive symptoms.
Change in Generalized Anxiety Disorder-7 (GAD-7) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  GAD-7 is a 7-item scale of general anxiety disorder that assesses anxiety symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 21. Higher scores indicate higher levels of anxiety.
Change in World Health Organization Disability Assessment Schedule (WHODAS 2.0) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  WHODAS 2.0 is a 12-item scale that measures ability to engage in daily activities. Each item is scored from 1 (none) to 5 (extreme) and ranges between 12 and 60. Higher scores indicate higher levels of daily dysfunctioning.
Change in Posttraumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual-5 (DSM-5) (PCL-5) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  PCL-5 is a 20-item questionnaire that assesses PTSD symptoms. Each item is scored from 0 (not at all) to 4 (extremely) providing a range between 0 and 80. Higher scores indicate higher levels of PTSD symptoms.
Change in Prolonged Grief Disorder-13 (PG-13) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  The PG-13 instrument contains 13 items: two items (items 3 and 13) on duration and impairment that are to be answered "yes" or "no", and 11 items assessing cognitive, behavioral and emotional symptoms, rated on a 5-point scale. Items 1, 2, 4 and 5 are rated on a frequency scale ranging from: "not at all" to "several times a day" (scoring 1-5), and items 6-12 are rated on an intensity scale ranging from "not at all" to "overwhelmingly" (scoring 1-5). These total scores, ranging from 11 to 55. Higher total scores on the PG-13 indicate more severe symptoms of prolonged grief.
Change in World Health Organization Quality of Life (WHOQOL-BREF) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  WHOQOL-BREF is a 26-item scale that measures quality of life. Each item is scored from 1 (not at all) to 5 (completely) providing a range between 26 and 130. Higher scores indicate higher levels of quality of life.
Change in Multidimensional Scale of Perceived Social Support (MSPSS) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  MSPSS is a 12-item scale that measures perceived social support. Each item is scored from 1 (very strongly disagree) to 7 (very strongly disagree) providing a range between 12 and 84. Higher scores indicate higher levels of perceived social support.
Change in World Health Organization-Five Well-Being Index (WHO-5) (1998) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  WHO-5 (1998) is a 5-item scale that measures well-being. Each item is scored from 0 (at no time) to 5 (all of the time) providing a range between 0 and 25. Higher scores indicate higher levels of well-being.
Change in Dispositional Hope Scale (DHS) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  DHS is a 12-item scale that measures dispositional hope. Each item is scored from 1 (definitely false) to 8 (definitely true) providing a range between 12 and 96. Higher scores indicate higher levels of dispositional hope.
Change in The Emotion Regulation Questionnaire (ERQ) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  ERQ is a 10-item questionnaire that measures emotion regulation. Each item is scored from 1 (strongly disagree) to 7 (strongly agree) providing a range between 10 and 70. Higher scores indicate higher levels of emotion regulation.
Change in Acceptance and Action Questionnaire - version 2 (AAQ-2) over time | Change from baseline assessment (one week before the first session of CA-CBT) to follow-up assessment (1 month after post-assessment)
  AAQ-2 is a 7-item questionnaire that measures of psychological inflexibility, experiential avoidance, and potential psychological distress. Each item is scored from 1 (never true) to 7 (always true) providing a range between 7 and 49. Higher scores indicate higher levels of psychological inflexibility, experiential avoidance, and more potential psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Şule N. Orhan, Study Chair — World Human Relief
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acarturk ZC, Abuhamdeh S, Jalal B, Unaldi N, Alyanak B, Cetinkaya M, Gulen B, Hinton D. Culturally adapted transdiagnostic CBT for SSRI resistant Turkish adolescents: A pilot study. Am J Orthopsychiatry. 2019;89(2):222-227. doi: 10.1037/ort0000310. Epub 2018 Jan 18. PMID 29345479
- [Background] Anadolu Agency. (2023c). Death toll from February earthquakes in Türkiye rises to 50,096. https://www.aa.com.tr/en/turkiye/death-toll-from-february-earthquakes-in-turkiye-rises-to-50-096/2850760
- [Background] Anik E, West RM, Cardno AG, Mir G. Culturally adapted psychotherapies for depressed adults: A systematic review and meta-analysis. J Affect Disord. 2021 Jan 1;278:296-310. doi: 10.1016/j.jad.2020.09.051. Epub 2020 Sep 15. PMID 32979561
- [Background] Bianchini V, Roncone R, Giusti L, Casacchia M, Cifone MG, Pollice R. PTSD Growth and Substance Abuse Among a College Student Community: Coping Strategies after 2009 L'aquila Earthquake. Clin Pract Epidemiol Ment Health. 2015 Mar 31;11:140-3. doi: 10.2174/1745017901511010140. eCollection 2015. PMID 25893001
- [Background] Bianchini V, Roncone R, Tomassini A, Necozione S, Cifone MG, Casacchia M, Pollice R. Cognitive behavioral therapy for young people after l'aquila earthquake. Clin Pract Epidemiol Ment Health. 2013 Nov 28;9:238-42. doi: 10.2174/1745017901309010238. eCollection 2013. PMID 24358053
- [Background] Cenat JM, McIntee SE, Blais-Rochette C. Symptoms of posttraumatic stress disorder, depression, anxiety and other mental health problems following the 2010 earthquake in Haiti: A systematic review and meta-analysis. J Affect Disord. 2020 Aug 1;273:55-85. doi: 10.1016/j.jad.2020.04.046. Epub 2020 May 7. PMID 32421623
- [Background] Chan CL, Wang CW, Ho AH, Qu ZY, Wang XY, Ran MS, Mao WJ, Lu BQ, Zhang BQ, Zhang XL. Symptoms of posttraumatic stress disorder and depression among bereaved and non-bereaved survivors following the 2008 Sichuan earthquake. J Anxiety Disord. 2012 Aug;26(6):673-9. doi: 10.1016/j.janxdis.2012.05.002. Epub 2012 May 29. PMID 22721751
- [Background] Ergun D, Senyuz S. Prolonged grief disorder among bereaved survivors after the 2011 Van Earthquake in Turkey. Death Stud. 2022;46(6):1364-1371. doi: 10.1080/07481187.2021.1884624. Epub 2021 Feb 12. PMID 33576723
- [Background] Farooqui M, Quadri SA, Suriya SS, Khan MA, Ovais M, Sohail Z, Shoaib S, Tohid H, Hassan M. Posttraumatic stress disorder: a serious post-earthquake complication. Trends Psychiatry Psychother. 2017 Apr-Jun;39(2):135-143. doi: 10.1590/2237-6089-2016-0029. PMID 28700042
- [Background] Geng F, Fan F, Mo L, Simandl I, Liu X. Sleep problems among adolescent survivors following the 2008 Wenchuan earthquake in China: a cohort study. J Clin Psychiatry. 2013 Jan;74(1):67-74. doi: 10.4088/JCP.12m07872. PMID 23419228
- [Background] Harada N, Shigemura J, Tanichi M, Kawaida K, Takahashi S, Yasukata F. Mental health and psychological impacts from the 2011 Great East Japan Earthquake Disaster: a systematic literature review. Disaster Mil Med. 2015 Sep 2;1:17. doi: 10.1186/s40696-015-0008-x. eCollection 2015. PMID 28265432
- [Background] Jiang S, Yan Z, Jing P, Li C, Zheng T, He J. Relationships between Sleep Problems and Psychiatric Comorbidities among China's Wenchuan Earthquake Survivors Remaining in Temporary Housing Camps. Front Psychol. 2016 Oct 18;7:1552. doi: 10.3389/fpsyg.2016.01552. eCollection 2016. PMID 27803679
- [Background] Lopes AP, Macedo TF, Coutinho ES, Figueira I, Ventura PR. Systematic review of the efficacy of cognitive-behavior therapy related treatments for victims of natural disasters: a worldwide problem. PLoS One. 2014 Oct 8;9(10):e109013. doi: 10.1371/journal.pone.0109013. eCollection 2014. PMID 25296020
- [Background] Orhan, Ş.N. (2020). Travma yaşayan kadınlara kültüre adapte edilmiş bilişsel davranışçı grup terapi uygulanması ve etkilerinin incelenmesi (Eng. The application of culturally adapted cognitive behavioral therapy and investigation of its impact in women with traumatic experiences). Unpublished master's thesis, Graduate School of Social Sciences, Marmara University, İstanbul.
- [Background] Shooshtary MH, Panaghi L, Moghadam JA. Outcome of cognitive behavioral therapy in adolescents after natural disaster. J Adolesc Health. 2008 May;42(5):466-72. doi: 10.1016/j.jadohealth.2007.09.011. Epub 2008 Mar 4. PMID 18407041
- [Background] Wen J, Shi YK, Li YP, Yuan P, Wang F. Quality of life, physical diseases, and psychological impairment among survivors 3 years after Wenchuan earthquake: a population based survey. PLoS One. 2012;7(8):e43081. doi: 10.1371/journal.pone.0043081. Epub 2012 Aug 21. PMID 22937014
- [Background] Yang CH, Xirasagar S, Chung HC, Huang YT, Lin HC. Suicide trends following the Taiwan earthquake of 1999: empirical evidence and policy implications. Acta Psychiatr Scand. 2005 Dec;112(6):442-8. doi: 10.1111/j.1600-0447.2005.00603.x. PMID 16279873
- [Background] Yi X, Gao J, Wu C, Bai D, Li Y, Tang N, Liu X. Prevalence and risk factors of prolonged grief disorder among bereaved survivors seven years after the Wenchuan earthquake in China: A cross-sectional study. Int J Nurs Sci. 2018 Apr 17;5(2):157-161. doi: 10.1016/j.ijnss.2018.04.001. eCollection 2018 Apr 10. PMID 31406818